CLINICAL TRIAL: NCT01608191
Title: Obesity Treatment With LCD(Low Calorie Diet) in Primary Health Care - Long Term Effects With or Without Internet Based CBT (Cognitive Behavioral Therapy) , for Weight Stability
Brief Title: Obesity Treatment With LCD in Primary Health Care
Acronym: LCD-KBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro County Council (Other Government)
Responsible Party: Principal Investigator, Jan Karlsson, Behaviorist, Örebro County Council
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCC-LCD-PV; 2011/434 (Other: Central Ethical Review Board, Uppsala Sweden)
Record Dates: First submitted 2012-05-25; First posted 2012-05-30 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Obesity; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ordinary primary care follow up (No Intervention): Ordinary follow up after 24 weeks of LCD diet + reintroduction of food.
- CBT follow up (Active Comparator): 11 weeks intervention programme with CBT conducted via internet.
  Interventions: Behavioral: CBT follow up

INTERVENTIONS:
Behavioral: CBT follow up — 11 weeks programme conducted via internet. CBT with focus on weight stability.
  Arms: CBT follow up

SUMMARY:
The aim of this study is to evaluate if an internet-based CBT (Cognitive Behavioral Therapy) programme for weight stability after LCD (Low Calorie diet) treatment for obesity, can reduce weight gain and improve weight stability, self reported health, pain, eating behavior, fatigue and mood.

Adults with obesity and health problems in primary health care are invited to be part of the study. The geographical area is Orebro county which has in all 29 primary health care centers. Population is 276 000, and according to population studies around 15% of the adult population has a BodyMassIndex (BMI) over 30, which is characterized as obesity according to WHO.

Specific objectives are;

* To evaluate if internet-based CBT treatment after LCD improves weight stability after 1 and 2 years.
* To evaluate if weight loss improves metabolic parameters such as HbA1c, blood glucose, Cholesterol, Low density lipoproteins (LDL),High density lipoproteins (HDL) , triglycerides (TG) and Bloodpressure (BP)
* To evaluate weight loss influence on quality of life, body pain, eating behavior, obesity related problems, fatigue and mood, and to see if CBT program for weight stability also improves these factors
* To evaluate if LCD treatment is a possible treatment for obesity in ordinary primary health care

Patients taking part in the study, undergo a 12 week period of Low Calorie Diet (LCD) treatment, followed by a 12 week reintroduction to ordinary food. During this period the patient has contact with the primary health care nurse and doctor. After 24 weeks of treatment, the patient who follows the study is supposed to have lost around 10% of initial weight.All patients losing more than 7% weight during the first 24 weeks, are randomized to either ordinary follow up (group 1) or an internet-based CBT programme for weight stability (group 2). All patients in the study are followed at 1 year by doctor, and at 2 year by nurse visit.

DETAILED DESCRIPTION:
Patients are recruited in an ordinary primary care setting in Primary care centers in Orebro County. All Primary care centers in the area (26) are invited to take part in the study.

Patients are given brief information at ordinary visits at doctor, nurse or physiotherapists, or by written information announced at the health care center. Before going into the study they need a doctors visit to pass the inclusion and exclusion criteria. The study starts at a nurse visit where the patient gets written information about the LCD treatment and the protocol.

After 24 weeks in the study, all patients with weight loss of 7% or more are randomized into two groups.

Group 1, keep their contact with the nurse at the primary health care centre, and gets a written prescription of physical activity, which is followed by a visit at 36 weeks.

Group 2, gets a code for the internet-based CBT programme. They go into the programme at home, and follow the programme which has the goal of weight stability and contains strategies of meal plans, portion controls, physical activity planning, and cognitive strategies of thinking and goal setting. During this programme there is an opportunity to "chat" with CBT therapists via the internet, concerning the programme and its challenges. No personal meeting with therapist is included.

At 1 year in the study both groups meed with doctor at primary health care center and at 2 year there is a nurse follow up at the same center.

At baseline, 12 weeks, 24 weeks, 1 year and 2 years several validated instruments are used to follow patients wellbeing due to:

* Quality of life (Short Form -36, SF-36)
* Obesity related problems (Obesity related Problems Scale version 3 OPv3)
* Mood (Mood Adjective Chek List MACL)
* Self reported pain (Brief Pain Inventory Short form BPI-SF)
* Eating behavior (Three Factor Eating Questionnaire- Revised 21 Items TFEQ-R21)
* Fatigue (Multidimensional Fatigue Inventory MFI)

We also investigate the patients experiences of the treatment, how they manage to hold on to the diet, and how it effects their motivation for ongoing lifestyle changes. For this we use a study specific instrument.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30 with health problems and willingness and motivation to make lifestyle changes.
* Access to the internet and the ability to read and understand written information in swedish.

Exclusion Criteria:

* BMI < 30
* Excessive eating disorder problems (screening forms are used)
* Severe heart failure (New York Heart Association (NYHA) class III-IV)
* Moderate or severe COPD (Chronic Obstructive Pulmonary Disease) (FEV% <50)
* Uncontrolled asthma (hospitalization or more than twice requiring inhalation treatment on health care site last year)
* Pregnancy and lactation
* Type 1 Diabetes
* Serious liver dysfunction (ALT value more than doubled, women> 1.5 μkat / L, men> 2.2 μkat / L)
* Former Gastric bypass surgery or other weight reducing surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
• Weight reduction in kg and % from baseline to 1 and 2 years | Change from baseline to follow up at 1 and 2 years
  Patients in the intervention group (Group 2) have an average of 5 kg greater weight loss at 1 year follow-up compared with patients in the control group (Group 1) Out of patients completing 1 year of treatment, 75% reached the weight loss -5%, and 50% have achieved weight loss - 10%

SECONDARY OUTCOMES:
• LCD treatment is an effective and suitable treatment for primary health care | Change from baseline to follow up at 1 and 2 years
  We use a questionnaire that states the patients view about the treatment, and also measurement of how many patients are lost to follow up, or do not go through the full treatment.
Improved metabolic control (lower weight and waist circumference, lower TGA) Higher HDL, lower Hba1c | From baseline to 1 year
  • Patients , regardless of treatment group, has improved metabolic control (higher HDL, lower TGA, lower weight and waist circumference) compared to baseline measurements at 1 year. Lower fasting plasma glucose (fP-glucose) and HbA1C in subgroup type 2 diabetics at 1 year compared to baseline.
Quality of life improvements in both groups compared with baseline at one year | baseline to 1 year
  • Quality of life and Obesity problems measured by SF36 and OPv3 improves with weight loss. Self reported pain (BPI-SF), eating behavior (TFEQ-R21), mood (MACL)and fatigue (MFI) also improves with weightloss in both groups.
  We also want to compare the two groups in order to see if the CBT programme has additional effects on these parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Karlsson, Principal Investigator — Universitetssjukvårdens forskningscentrum, UFC, Region Örebro län, Box 1613, 70116 Örebro
Locations (1):
- Orebro County Council, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No